CLINICAL TRIAL: NCT05428774
Title: Efficacy of Different Oral Rehydration Solutions on the Hydration Status of Healthy Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liquid I.V. (Other)
Collaborators: Lipscomb University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Pilot
Record Dates: First submitted 2022-06-15; First posted 2022-06-23 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Fluid Retention; Beverage Hydration Index; Hydration Status

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test Product 1 (Experimental): Participants will consume test product 1 during one experimental visit.
  Interventions: Other: Test product 1
- Test Product 2 (Experimental): Participants will consume test product 2 during one experimental visit.
  Interventions: Other: Test product 2
- Placebo (Placebo Comparator): Participants will consume placebo during one experimental visit.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Test product 1 — Participants will receive TP1 during one experimental visit.
  Arms: Test Product 1
Other: Test product 2 — Participants will receive TP2 during one experimental visit.
  Arms: Test Product 2
Other: Placebo — Participants will receive placebo during one experimental visit.
  Arms: Placebo

SUMMARY:
Dehydration lowers both physical and mental performance if it is severe enough. Performance declines are more pronounced in hot conditions or after prolonged strenuous activity such as exercise. Most individuals drink less than their sweat losses during activity, while some individuals overdrink and develop a sodium deficiency. Water and electrolyte balance must be restored as part of the recovery process after any activity that causes sweating. Plain water causes a decrease in plasma sodium concentration and osmolality, which reduces the desire to drink and increases urine production. Unless the volume ingested exceeds the loss, individuals are in net negative fluid balance throughout the recovery period due to urinary losses. When sodium and potassium are added to rehydration fluids, urine production is reduced in the hours following rehydration. Rehydration is only possible if a volume of fluid equal to or greater than the amount lost through sweat is consumed, together with adequate electrolytes. The two test products for this study, are novel hydration beverage formulas. They are an electrolyte drink mixture with five essential vitamins and three times more electrolytes than typical sports beverages. The test products create an osmotic force that permits water to be supplied to the bloodstream sooner in the digestive system by using a specific ratio of sodium, glucose, and potassium. This randomized, placebo-controlled, semi-blind, crossover study will evaluate the effects of the test products on rehydration in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males 18-35 years old at the time of screening. Participants need to be competent i.e., able to understand what is to take place and able to provide a free decision on agreeing to the activity/taking part in the study. Participants must be able to read and understand study instructions and any other relevant study documents. Willing to following the lifestyle and dietary restrictions as detailed in the Information Sheet for study.

Exclusion Criteria:

* A history or presence of a clinically relevant cardiac, renal, hepatic, endocrine (including diabetes mellitus), pulmonary, biliary, gastrointestinal, pancreatic, or neurologic disorder. Consumption other nutritional supplements, performance enhancing drugs, and non-steroidal anti-inflammatory drugs (NSAIDs) during the clinical. Participant has any medical condition which alters fluid balance in the body as confirmed by a health history questionnaire. Following a dietary pattern which may alter our findings (e.g., low carbohydrate/ketogenic diet, carnivore diet, intermittent fasting etc.). Women are excluded due to the variability of fluid retention during the menstrual cycle. Participant is not currently enrolled in another clinical study. Participant is consuming any medication which may alter fluid retention such as diuretics. The participant is an employee of the Sponsor.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Beverage hydration index | Through study completion, average of 6 weeks
  The primary objective of this study is to investigate the efficacy of two different oral rehydration solutions on the hydration status in healthy males via the beverage hydration index
Hydration status | Through study completion, average of 6 weeks
  The primary objective of this study is to investigate the efficacy of two different oral rehydration solutions on the hydration status in healthy males via urine specific gravity analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Townsend, PhD, Principal Investigator — Lipscomb University
Locations (1):
- Lipscomb University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No